CLINICAL TRIAL: NCT03581669
Title: Acetabular Cerclage and Total Hip Arthroplasty in the Treatment of Acetabular Fractures in Elderly Patients.
Acronym: jantjeVL
Status: Withdrawn | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: BJCerTHA; UZ leuven (Other: UZ leuven)
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Elderly; Acetabular Fractures; Cerclage Acetabular Fractures; Total Hip Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — cerclage and THA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- THA + cerclage acetabulum
  Interventions: Device: Cerclage and total hip arthroplasty

INTERVENTIONS:
Device: Cerclage and total hip arthroplasty — acetabular fractures in the elderly treated with cerclage acetabulum and total hip arthroplasty

SUMMARY:
We want to present the outcome of complex multifragmented acetabular fractures in the elderly treated with acetabular cerclage and total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* elderly (>60Years)
* acetabular fracture

Exclusion Criteria:

* Revision surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: elderly patients who sustained an acetabular fracture
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-08 (Estimated); Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
harris hip score | 1 year
  outcome after cerclage and THA

CONTACTS AND LOCATIONS:
Overall Officials: Vanderschot Paul, MD, Phd, Principal Investigator — UZ Leuven; Molenaers Guy, MD, Phd, Study Chair — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Background] Mouhsine E, Garofalo R, Borens O, Blanc CH, Wettstein M, Leyvraz PF. Cable fixation and early total hip arthroplasty in the treatment of acetabular fractures in elderly patients. J Arthroplasty. 2004 Apr;19(3):344-8. doi: 10.1016/j.arth.2003.08.020. PMID 15067649